CLINICAL TRIAL: NCT03677999
Title: Spectroscopic Magnetic Resonance Imaging of Glioma
Acronym: MEGA-PRESS
Status: Withdrawn | Type: Observational
Why Stopped: Faculty left the institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUROSURG-2018-26848
Record Dates: First submitted 2018-09-13; First posted 2018-09-19 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor-Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brain tumor patients with Glioma: 1. Men and women scheduled who are diagnosed with glioma who is seeking clinical care for their conditions at the UMN Masonic cancer center.
  2. Passed the safety screen for MRI
  3. Age 18 or older Participants will receive MEGA-PRESS sequence Magnetic Resonance Spectroscopy during their routined schedule standard of care MRI.
  Interventions: Diagnostic Test: MEGA-PRESS sequence Magnetic Resonance Spectroscopy

INTERVENTIONS:
Diagnostic Test: MEGA-PRESS sequence Magnetic Resonance Spectroscopy — MRS protocols and novel MRI methods that allow detection and quantification of 2 hydroxyglutarates (2HG) as well as the physiologic consequences of 2HG accumulation.

SUMMARY:
The study is designed to develop and test new Magnetic Resonance Imaging methods that can improve the characterization of brain cancer and facilitate improved clinical care of these participants.

DETAILED DESCRIPTION:
The primary objective of this study is to develop and test new Magnetic Resonance Imaging methods that can improve the characterization of brain cancer and facilitate improved clinical care of these participants. More specifically, investigators are interested in applying novel spectroscopic and quantitative MR methods that give information beyond what is produced by a clinical brain MRI study and to understand the clinical correlates of the imaging findings. Investigators have tested these sequences in healthy volunteers. The investigators now wish to test these sequences in brain cancer participants in order to understand how these sequences can best be applied in a clinical setting.

To acquire these data, investigators intend to perform additional MRI acquisitions on participants who are scheduled to receive a clinical MRI at the UMN Center for Clinical Imaging Research (CCIR), a facility located at the Center for Magnetic Resonance Research (CMRR). Since these MRIs are required for the participants' clinical care, the participant will not be making additional visits to the CCIR. Based on published data and pilot experiences reported from other institutions, the sequences are well-tolerated. The only imposition for the participant is that the participant will spend additional time in the scanner after completion of the imaging required for clinical care. An informed consent form describing the additional MR sequences performed will be presented to the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women scheduled who are diagnosed with glioma who is seeking clinical care for their conditions at the UMN Masonic cancer center.
2. Passed the safety screen for MRI
3. Age 18 or older
4. Ability to read and understand English
5. Ability to provide informed consent

Exclusion Criteria:

1. Participants who are excluded from the base MRI scan, as determined by the CMRR/CCIR clinical policies are necessarily excluded from this study, as the MRI scan will not be performed.
2. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Glioma who is seeking clinical care for their conditions at the UMN Masonic cancer center Aand scheduled to have standard of care MRI.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2024-09-14 (Estimated); Study Completion 2025-09-14 (Estimated)

PRIMARY OUTCOMES:
The number of brain cancer participants with IDH mutation status | 30 minutes
  MEGA-PRESS MRI sequence will be utilized to determine IDH status

CONTACTS AND LOCATIONS:
Overall Officials: Clark Chen, MD, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data may be shared with other investigators via a web-based University of Minnesota Box secured storage. Box Secure Storage is a secure environment delivered by the Center of Excellence for HIPAA Data intended for storing, sharing and accessing sensitive and private-highly restricted files.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 2 years
Access Criteria: The link to the data will be made available upon request